CLINICAL TRIAL: NCT06625138
Title: Single-blinded Randomized Trial of Latex Vs Non-latex Hemorrhoid Banding
Brief Title: Trial of Latex Vs Non-latex Hemorrhoid Banding
Acronym: NO-Tex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huntington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Adam Truong, Investigator, Huntington Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY0003511
Record Dates: First submitted 2024-09-11; First posted 2024-10-03 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hemorrhoid; Hemorrhoid Bleeding
Keywords: hemorrhoid; banding
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non-latex band (Experimental): Non-latex bands will be placed on hemorrhoids during banding
  Interventions: Device: Non-Latex Band
- Latex band (Active Comparator): latex bands will be placed on hemorrhoids during banding
  Interventions: Device: Latex Band

INTERVENTIONS:
Device: Latex Band — Hemorrhoid banding with latex band
  Arms: Latex band
Device: Non-Latex Band — Hemorrhoid banding with non-latex bands
  Arms: Non-latex band

SUMMARY:
This study will involve the recruitment of adult patients with hemorrhoids for whom rubber band ligation is the recommended treatment. Patients will be randomized to receive banding with a latex band or non-latex band. Our goal will be to measure the performance of latex bands vs non-latex bands.

DETAILED DESCRIPTION:
This study will involve the recruitment of adult patients with symptomatic grade 2-3 internal hemorrhoids for whom rubber band ligation is the recommended treatment. Patients will be randomized to receive banding with a latex band or non-latex band. Our hypothesis is that non-latex hemorrhoidal bands are non-inferior to latex bands for the treatment of grade 2-3 internal hemorrhoids.

The secondary objective of the study is to compare banding-related adverse effects including pain, bleeding, and complications assessed both immediately and within 3 weeks following each hemorrhoidal banding.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade 2-3 internal hemorrhoids undergoing rubber band ligation

Exclusion Criteria:

* Previous hemorrhoidal banding within the past year
* Known latex allergy
* Pregnancy
* Anticoagulation use
* Bleeding disorder
* Portal hypertension
* Inflammatory bowel disease
* Immunosuppression
* Functional neurologic disorder
* Pelvic floor dysfunction
* Any records flagged "break the glass" or "research opt out".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Hemorrhoid Band Efficacy | 2-4 months
  hemorrhoidal bleeding and prolapse symptoms following ligation.

SECONDARY OUTCOMES:
Banding-related Adverse events | 2-4 months
  banding-related adverse events including pain, bleeding, and complications following hemorrhoidal banding

CONTACTS AND LOCATIONS:
Overall Officials: Adam Truong, MD, Principal Investigator — Huntington Health
Locations (1):
- Huntington Memorial Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from start of study for 2 years
Access Criteria: Data will be available upon reasonable request